CLINICAL TRIAL: NCT01685788
Title: Prospective Longitudinal Study: Sensory Deficits in the Upper Limb After Stroke.
Brief Title: Study of Sensory Deficits in the Upper Limb After Stroke
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Sarah Meyer, PhD Student, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: KUL - FaBeR - Stroke - Meyer
Record Dates: First submitted 2012-09-06; First posted 2012-09-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- study participants
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The overall aim of the project is to gain insight in sensory deficits and recovery patterns in the upper limb post stroke and its association with brain lesion localisation. Furthermore, the investigators will identify associations of deficits in sensory modalities with upper limb impairments, activities and participation at different time points after stroke. Identification of the sensory deficits, along with further insights in their relation with objective neurophysiological and neuroanatomical measures will contribute to the amelioration of goal-setting for the rehabilitation of upper extremity function after stroke. These functions are indispensable during several daily activities as well in different sports and leisure activities. This project is an important step towards a better delineating of treatment interventions for the upper limb and to a better guiding of individual needs for post-stroke treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* first-ever stroke as defined by WHO
* ≤ 5 days post stroke
* motor impairment and/or a sensory impairment
* ≥ 18 years old
* sufficient cooperation to execute evaluations

Exclusion Criteria:

* other neurological impairments such as previous stroke, head injury or multiple sclerosis (these might affect sensory ability independently of the stroke)
* stroke-like symptoms caused by subdural hematoma, tumour, encephalitis or trauma
* no informed consent
* pre-stroke Barthel Index < 95 out of 100 points (to be able to distinguish between pre-existing disabilities and disabilities resulting from the stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in sensory function in upper limb from baseline up to 6 months post stroke | 6 months post stroke

SECONDARY OUTCOMES:
Change in motor function in upper limb from baseline up to 6 months post stroke | 6 months post stroke

OTHER OUTCOMES:
activity measure | 6 months post stroke
  The investigators will use the ABILHAND Questionnaire, a measure of how well the hemiplegic arm and hand can be used in daily activities.
Activity measure | 6 months after stroke
  The Assisting Hand Assessment (AHA) will be used to investigate the use of the hemiplegic arm in bimanual tasks after stroke.
Participation measure | 6 months after stroke
  The quality of life will be measured using the Stroke Impact Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Professor, Principal Investigator — Catholic University Leuven; Sarah Meyer, PhD student, Principal Investigator — Catholic University Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium